CLINICAL TRIAL: NCT02273505
Title: Comparison of Pharmacokinetics of Dipyridamole in Asasantin Extended Release (ER) 200/25 mg Capsules Bid and in a Combination of Persantin Immediate Release Tablets (100 mg Qid) and ASA Tablets (25 mg Bid) in an Open, Randomized, 2-way Crossover Study in Healthy Subjects
Brief Title: Comparison of Pharmacokinetics of Dipyridamole in Asasantin Extended Release (ER) and in a Combination of Persantin Immediate Release Tablets and ASA Tablets in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 9.138
Record Dates: First submitted 2014-10-23; First posted 2014-10-24 (Estimated); Last update posted 2014-10-24 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
MeSH Terms: interventions — Aspirin, Dipyridamole Drug Combination; Dipyridamole

ARMS (2):
- Asasantin (ER) (Experimental)
  Interventions: Drug: Asasantin (ER)
- Combination of Persantin and ASA (Active Comparator)
  Interventions: Drug: Persantin; Drug: Acetyl salicylic acid (ASA)

INTERVENTIONS:
Drug: Asasantin (ER)
  Arms: Asasantin (ER)
Drug: Persantin
  Arms: Combination of Persantin and ASA
Drug: Acetyl salicylic acid (ASA)
  Arms: Combination of Persantin and ASA

SUMMARY:
Comparative Pharmacokinetics of Asasantin Extended Release (ER) and of immediate release Persantin tablets combined with Acetyl salicylic acid (ASA) tablets

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects as determined by results of screening
* Signed informed consent in accordance with Good Clinical Practice (GCP) and local legislation
* Age >= 18 and <= 55 years
* Broca >= - 20% and <= + 20%

Exclusion Criteria:

* Any findings of the medical examination (including blood pressure, pulse rate and ECG) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorder
* Surgery of the gastro-intestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* Chronic or relevant acute infections
* History or hypersensitivity to Asasantin ER and any of the excipients
* Intake of drugs with a long half-life (> 24 hours) (<= 1 month prior to administration or during the trial)
* Use of any drugs which might influence the result of the trial (<= 10 days prior to administration or during the trial)
* Participation in another trial with an investigational drug (<= 1 month prior to administration or during the trial)
* Known alcohol abuse
* Known drug abuse
* Blood donation ( <=1 month prior to administration or during the trial)
* Excessive physical activities (<=5 days prior to administration or during the trial)
* History of hemorrhagic diseases
* History of gastro-intestinal ulcer, perforation or bleeding
* History of bronchial asthma
* Any laboratory value outside the reference range of clinical relevance

For female subjects:

* Pregnancy
* Positive pregnant test
* No adequate contraception (adequate contraception e.g. sterilization, intrauterine device (IUD), oral contraceptives)
* Inability to maintain this adequate contraception during the whole study period
* Lactation period

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2000-04; Primary Completion 2000-05 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve at steady state (AUCss) | Up to 144 hours after drug administration
Percentage peak trough fluctuation (%PTF) | Up to 144 hours after drug administration

SECONDARY OUTCOMES:
Maximum plasma concentration at steady state (Cmax,ss) of dipyridamole (dp) | Up to 144 hours after drug administration
Maximum plasma concentration at steady state / Area under the plasma concentration-time curve at steady state ((Cmax,ss) / (AUCss)) of dipyridamole | Up to 144 hours after drug administration
Time to reach maximum plasma concentration at steady state (tmax,ss) of dipyridamole | Up to 144 hours after drug administration
Fluctuation of AUC (AUCfluct) of dipyridamole | Up to 144 hours after drug administration
Terminal half-life in the analyte (t1/2) of dipyridamole | Up to 144 hours after drug administration
Urinary excretion (Ae%) of dp, dipyridamole glucuronide (dp-gluc) and salicylic acid (SA) | Up to 106 hours after drug administration
Number of participants with abnormal changes in clinical laboratory parameters | Up to day 7 after last drug administration
Number of participants with Adverse Events | Up to day 7 after last drug administration